CLINICAL TRIAL: NCT06707337
Title: The Effects of a Brief Self-compassion Program Applied to Patients With Colorectal Cancer on Self-compassion and Self-care
Brief Title: Brief Self-Compassion Program in Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kübra DAKDEVİR (Other Government)
Collaborators: Çankırı Karatekin University (Other)
Responsible Party: Sponsor-Investigator, Kübra DAKDEVİR, Nurse, Ankara Etlik City Hospital
Organization: Ankara Etlik City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ankara Etlik Şehir Hastanesi
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer
Keywords: Cancer; Self-Compassion; Self-care; Colorectal Cancer; Randomized Controlled Trial
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: The study was planned as a prospective, two-armed (1:1), randomized controlled experimental study. This randomized controlled trial will be reported according to the CONSORT guidelines.
Who Masked: Participant
Masking Description: Patients with colorectal cancer in the experimental and control groups will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participant Group (Experimental): Brief Self-compassion Program will be held in a face-to-face hospital environment for the patients with colorectal cancer in the experimental group. This training program has been developed based on the concepts of Mindfulness-Based Compassionate Living and Mindfulness-Based Stress Reduction Programs. The content and topics of the sessions in the program are arranged according to the conceptual structure and flow of the mindfulness-based model. The training program was created in a certain flow, based on the introduction to a short self-compassion program (1 sessions), the importance of self-compassion and self-care in the cancer experience (1 sessions), a self-compassionate approach to challenging emotions and situations (1 sessions). There are 3 sessions in the program and the frequency of sessions is 3 times a week, and each session lasts approximately 45 minutes. The training program will be applied to 33 patients with colorectal cancer in the experimental group.
  Interventions: Other: Brief Self-compassion Program
- Control Group (No Intervention): There will be no training or intervention.

INTERVENTIONS:
Other: Brief Self-compassion Program — Brief Self-compassion Program will be held in a face-to-face hospital environment for the patients with colorectal cancer in the experimental group. This training program has been developed based on the concepts of Mindfulness-Based Compassionate Living and Mindfulness-Based Stress Reduction Programs. The content and topics of the sessions in the program are arranged according to the conceptual structure and flow of the mindfulness-based model. The training program was created in a certain flow, based on the introduction to a short self-compassion program (1 sessions), the importance of self-compassion and self-care in the cancer experience (1 sessions), a self-compassionate approach to challenging emotions and situations (1 sessions). There are 3 sessions in the program and the frequency of sessions is 3 times a week, and each session lasts approximately 45 minutes. The training program will be applied to 33 patients with colorectal cancer in the experimental group.
  Arms: Participant Group

SUMMARY:
In this study, between 1 December 2024-31 March 2025, who met the inclusion and exclusion criteria, a total of 66 patients with colorectal cancer at the Etlik City Hospital General Surgery Department.

DETAILED DESCRIPTION:
Brief Self-compassion Program will be held in a face-to-face hospital environment for the patients with colorectal cancer in the experimental group. This training program has been developed based on the concepts of Mindfulness-Based Compassionate Living and Mindfulness-Based Stress Reduction Programs. The content and topics of the sessions in the program are arranged according to the conceptual structure and flow of the mindfulness-based model. The training program was created in a certain flow, based on the introduction to a short self-compassion program (1 sessions), the importance of self-compassion and self-care in the cancer experience (1 sessions), a self-compassionate approach to challenging emotions and situations (1 sessions). There are 3 sessions in the program and the frequency of sessions is 3 times a week, and each session lasts approximately 45 minutes. The training program will be applied to 33 patients with colorectal cancer in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Can speak and understand Turkish
* Has written permission
* Being hospitalized in the General Surgery Clinic of the relevant institution on the dates of the study
* Diagnosed with colorectal cancer
* Having no mental illness that would prevent participation in the study

Exclusion Criteria:

* Not knowing the diagnosis
* Receiving or having received any psychosocial support or training
* Having previously participated in programs related to self-compassion
* Being meditating
* Having any history of mental retardation or organic brain damage that would prevent participation in the training
* Having a problem with understanding and following the given instructions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Self-Compassion Scale | Change from before implementation, after practice is completed (1th week)
  In order to determine the self-compassion levels of the patients participating in the study, the Self-Compassion Scale, which was developed by Neff (2003) (Neff, 2003) and adapted to Turkish by Akın, Akın and Abacı (2007) (Akın et al., 2007), was used. The English form of the Self-Compassion Scale consists of 26 items and 6 subscales. These subscales are self-compassion, isolation, awareness of sharing, self-judgment, over-identification and mindfulness. The self-kindness sub-dimension includes items 2, 6, 13, 17, 21, the self-judgment sub-dimension includes items 4, 7, 15, 20, 26, the awareness of sharing sub-dimension includes items 1, 8, 12, 22, the isolation sub-dimension includes items 5, 11, 19, 25, the conscious awareness sub-dimension includes items 9, 14, 18, 23, and the over-identification sub-dimension includes items 3, 10, 16, 24. The scale is a 5-point Likert-type scale with the ratings "1 Never", "2 Rarely", "3 Often", "4 Usually", "5 Always". The factor loadings in all
Mindful Self-Care Scale (MSCS) | Change from before implementation, after practice is completed (1th week)
  The scale, developed by Cook-Cottone and Guyker in 2018, consists of 33 items covering self-care behaviors (Cook-Cottone and Guyker, 2018). The scale consists of 5-point Likert-type questions and only the 6th item is reverse coded. The sub-dimensions of the scale consist of physical care, supportive relationships, conscious awareness, self-compassion and purpose, conscious relaxation, and supportive structure. As the scores obtained from the scale increase, it is seen that the individual's self-care skills are high. The internal consistency coefficient of the scale was found to be 0.89 overall, 0.69 for physical care, 0.86 for supportive relationships, 0.92 for awareness, 0.83 for self-compassion and purpose, 0.77 for conscious relaxation, and 0.77 for the supportive structure subscales. The scale was adapted to Turkish by Aydın Sünbül and colleagues in 2018 (Aydın Sünbül et al., 2018). After adaptation to Turkish, the scale maintained its subdimensions, while the internal consistency

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)